CLINICAL TRIAL: NCT02076490
Title: The PACT Trial - PAtient Centered Telerehabilitation: Effectiveness of Software-supported and Traditional Mirror Therapy in Patients With Phantom Limb Pain Following Lower Limb Amputation: Design of a Randomized Controlled Trial.
Brief Title: Telerehabilitation Using Mirror Therapy in Patients With Phantom Limb Pain Following Lower Limb Amputation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zuyd University of Applied Sciences (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 005-GW02-035
Record Dates: First submitted 2014-02-03; First posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Phantom Limb Pain
Keywords: Telerehabilitation, mirror therapy, phantom limb pain
MeSH Terms: conditions — Phantom Limb | interventions — Restraint, Physical; Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Software Supported Mirror Therapy (Experimental): First experimental condition Physical/Occupational Therapy
  Interventions: Other: Physical/Occupational therapy
- Traditional mirror therapy (Experimental): Second experimental condition Physical/Occupational Therapy
  Interventions: Other: Physical/Occupational therapy
- Sensomotor exercises without mirror (Active Comparator): Control condition Physical/Occupational Therapy
  Interventions: Other: Physical/Occupational therapy

INTERVENTIONS:
Other: Physical/Occupational therapy — At least 10 individual sessions over the clinical intervention period of 4 weeks followed by a 6 weeks self-management phase.

SUMMARY:
The overall aim of this randomized controlled study is to investigate the effectiveness of mirror therapy supported by telerehabilitation on the intensity, duration and frequency of phantom limb pain and daily activities compared to traditional mirror therapy and sensomotor exercises without a mirror in patients following lower limb amputation.

DETAILED DESCRIPTION:
Up to 75% of patients after amputation of an arm or leg suffer from chronic phantom limb pain that still is perceived in the missing limb, leading to limitations in daily activities and quality of life. The treatment of phantom limb pain is still challenging. Despite many different pharmacological interventions, the outcomes on the longer-term are in many cases not satisfying. Alternative, non-pharmacological interventions, such as mirror therapy, are gaining increased recognition in the treatment of phantom limb pain. In this context, telerehabilitation plays an important role to support long-term self-management and autonomy of these patients.

In the developmental phase of the project, a user-centred design is applied. Patients as well as physical and occupational therapists are interviewed concerning their preferences and needs with respect to the design and content of the telerehabilitation. Additionally, two focus groups with each five participants will be conducted. Subsequently, a prototype of the telerehabilitation will be developed based on user preferences, available evidence, expert opinion and already existing systems. This prototype will be tested on its usability and technical performance in phase three using the thinking-aloud-method and data logging. Accordingly, a multicenter, randomized controlled trial will be conducted to evaluate the cost-effectiveness of the telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Lower limb amputation
2. At least since one week constant or intermittent phantom limb pain (PLP) with an average intensity of at least score 3 on the 11-point NRS and a minimum frequency of one episode of PLP per week.
3. Sufficient cognitive, communicative and motor functions to be able to use the telerehabilitation service, to concentrate for at least 15 minutes on the mirror image and to follow instructions and questionnaires; this is based on clinical judgment of recruiting physicians or therapists.

   Exclusion Criteria:
4. Duration of inpatient rehabilitation not long enough to ensure the 4-week clinical intervention phase.
5. Bilateral amputation, severe co-morbidity (e.g. stroke) or pain affecting the intact limb; this prevents engagement in the prescribed exercise programs of the study.
6. Severe psychiatric disorders that preclude patients from participating in the trial.
7. Intensive course of mirror therapy in the past (> 6 treatments during the last three months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in average intensity of phantom limb pain | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: 11-point NRS
Change in frequency of phantom limb pain | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
Change in duration of phantom limb pain | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up

SECONDARY OUTCOMES:
Change in pain related limitations in daily activities | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: PDI, PSFS
Change in pain specific self-efficacy | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: Pain specific self-efficacy scale
Change in quality of life | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: EQ-5D-5L
Change in global perceived effect | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: GPE scale
Change in dimensions of phantom limb pain | At baseline, 4 and 6 weeks following baseline and at 6 months follow-up
  Measurement instrument: Neuropathic Pain Symptom Inventory (NPSI)

CONTACTS AND LOCATIONS:
Overall Officials: Rob J Smeets, Prof., Dr., Study Director — Research School CAPHRI, Maastricht University, Maastricht, The Netherlands

REFERENCES:
- [Derived] Rothgangel AS, Braun S, Schulz RJ, Kraemer M, de Witte L, Beurskens A, Smeets RJ. The PACT trial: PAtient Centered Telerehabilitation: effectiveness of software-supported and traditional mirror therapy in patients with phantom limb pain following lower limb amputation: protocol of a multicentre randomised controlled trial. J Physiother. 2015 Jan;61(1):42; discussion 42. doi: 10.1016/j.jphys.2014.08.006. Epub 2014 Oct 16. PMID 25439709